CLINICAL TRIAL: NCT02320994
Title: Managing Aftercare for Stroke (MAS): MAS-I - a Cross Sectional Study of Post-rehabilitation Stroke Burden and Patients' Needs
Acronym: MAS-I
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Prof. Dr. Ian Wellwood (Unknown); Prof. Dr. Jörg Wissel (Unknown); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: MAS-I
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Ischemic Stroke
Keywords: stroke; aftercare
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stroke patients: post-rehabilitation stroke patients

SUMMARY:
In this first step of the study the investigators will assess the needs, disease burden and current treatments of long-term stroke patients (phase MAS-I).

The ultimate aim of the complete MAS project (MAS I, II & III) is the development of a model of stroke aftercare delivery that can be evaluated to estimate effects in both our local and the wider stroke population.

DETAILED DESCRIPTION:
After discharge from hospital the current healthcare system in Germany allows considerable flexibility (therefore complexity) of patient access and mobility between multiple care providers in the community setting. The investigators believe this aftercare could be better coordinated by a specialized coordinated stroke aftercare service. Comprehensive coordinated multidisciplinary care is a proven concept with proven benefits in both acute and rehabilitation care provided in stroke units and neurorehabilitation centres. In this study the investigators postulate that a similar coordinated approach to care can be extended to the phase after in-patient rehabilitation has ended (i.e. "long-term management" as opposed to "early supported discharge") for disabled patients with stroke living in the community.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Participation in one of the previously conducted stroke cohort studies: STRAWINSKI or PREDICT
* Modified Rankin Score (mRS) recorded as = 1 - 5 (at last follow up during cohort study)
* Informed consent signed by patient or legal representative

Exclusion Criteria:

* Unwilling to have pseudonymised data stored, analyzed & anonymously published.
* Patients participating in the previous studies recruited in centres outside Berlin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in long term course after a moderate to severe ischemic stroke
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of unmet Needs | once
  Unmet needs of patients and carers after discharge from Rehabilitation. Score of variables examined (self-reported stroke related need, post-stroke spasticity, post-stroke pain, post-stroke aphasia, neuropsychological impairment, post-stroke depression, post-stroke dementia, inadequate secondary prevention, social care need and carer burden).

SECONDARY OUTCOMES:
post-stroke checklist | once
  Evaluation of post-stroke checklist as a valid tool to screen for relevant burden of disease after stroke.
Standard practice evaluation | once
  Comparison of Standard practice in relation to evidence-based recommendations and current Clinical Guidelines for the management of stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charité - Universitätsmedizin Berlin, NeuroCure Clinical Research Center & Center for Stroke Research Berlin; Ian Wellwood, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, Center for Stroke Research Berlin (CSB); Jörg Wissel, Prof. Dr., Principal Investigator — Neurologie und Psychosomatik am Wittenbergplatz
Locations (1):
- Charité - Universitätsmedizin Berlin (Center for Stroke Research Berlin CSB & NeuroCure Clinical Research Center), Berlin, Germany

REFERENCES:
- [Result] Hotter B, Padberg I, Liebenau A, Knispel P, Heel S, Steube D, Wissel J, Wellwood I, Meisel A. Identifying unmet needs in long-term stroke care using in-depth assessment and the Post-Stroke Checklist - The Managing Aftercare for Stroke (MAS-I) study. Eur Stroke J. 2018 Sep;3(3):237-245. doi: 10.1177/2396987318771174. Epub 2018 Apr 19. PMID 31008354
- [Result] Lehnerer S, Hotter B, Padberg I, Knispel P, Remstedt D, Liebenau A, Grittner U, Wellwood I, Meisel A; BSA Long Term Care Study Group. Social work support and unmet social needs in life after stroke: a cross-sectional exploratory study. BMC Neurol. 2019 Sep 6;19(1):220. doi: 10.1186/s12883-019-1451-y. PMID 31492151
- [Result] Padberg I, Hotter B, Liebenau A, Knispel P, Lehnerer S, Heel S, Wellwood I, Meisel A. Unmet Need for Social and Emotional Support and Lack of Recalled Screening Is Associated with Depression in the Long-Term Course After Stroke. Risk Manag Healthc Policy. 2020 Apr 1;13:285-293. doi: 10.2147/RMHP.S228265. eCollection 2020. PMID 32280291